CLINICAL TRIAL: NCT00179166
Title: Assessment of Metabolic Response in Critically Ill Patients With Acute Renal Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Vanderbilt University (Other)
Responsible Party: Alp Ikizler, MD, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30941
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Acute Renal Failure
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): supplement contains protein content of 1.4 g/kg/day
  Interventions: Drug: TPN nutritional supplement
- 2 (Active Comparator): supplement contains protein content of 2.0 g/kg/day
  Interventions: Drug: TPN nutritional supplement

INTERVENTIONS:
Drug: TPN nutritional supplement — intravenous administration of nutritional supplement for 4 hours at a dosage of 30 kcal/kg/day, in the form of lipids, carbohydrates and protein; the non-protein calories are comprised of lipids (30%) and carbohydrates (70%)

SUMMARY:
We hypothesize that a nutritional supplementation with higher than standard protein content (2.0 gm/Kg/day vs 1.4 gm/Kg/day) will result in improved whole-body net protein balance when administered to critically ill patients with acute renal failure (ARF).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age admitted to the intensive care unit
* New onset acute renal failure (ARF) or ARF superimposed on chronic kidney disease
* ARF will be defined by a sustained (over 24 hours) increase in serum creatinine > 0.5 mg/dl from baseline
* Patients will be recruited for the study within 3-5 days following establishment of ARF

Exclusion Criteria:

* Institutionalized patient
* Previous kidney transplant
* Pregnancy
* Unable to obtain consent from subject or legally recognized representative
* ARF from urinary tract obstruction or a volume responsive pre-renal state.
* Liver Failure
* Recent cerebrovascular accident (CVA)
* Coagulopathy defined as: Platelets < 50, PT > 20, INR > 2.0 if the patient requires the placement of an arterial or venous catheter; if the patient does not require the placement of an arterial or venous catheter for the study, coagulopathy will not be a basis for exclusion.
* Life expectancy < 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-06; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
whole-body net protein balance | 10 hours

SECONDARY OUTCOMES:
Net skeletal muscle protein balance | 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States